CLINICAL TRIAL: NCT04213469
Title: a Safety and Efficacy Evaluation of PD1-CD19-CART in Patients With Relapse/Refractory B-cell Lymphoma
Brief Title: PD1-CD19-CART in Patients With r/r B-cell Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioray Laboratories (Industry)
Collaborators: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019-CAR-00CH1
Record Dates: First submitted 2019-12-26; First posted 2019-12-30 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: Patients will receive one of the three doses of 2*10^6/kg, 4*10^6/kg,6*10^6/kg.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD1-CD19-CART (Experimental): Patients undergo leukapheresis. Patients will receive a lymphodepletion chemotherapy with cyclophosphamide and fludarabine before CART infusion. A dose of PD1-CD19-CART will be infused on day 0.
  Interventions: Biological: PD1 specific integrated anti-CD19 Chimeric Antigen Receptor T Cells

INTERVENTIONS:
Biological: PD1 specific integrated anti-CD19 Chimeric Antigen Receptor T Cells — Gene editing autologous T cells with anti-CD19 ScFv expression and knockout of PD1
  Other Names: PD1-CD19-CART

SUMMARY:
This is an open label, single-site, dose-escalation study in up to 25 participants with relapse/refractory B-NHL. This study aims to evaluate the safety and efficacy of the treatment with PD1-CD19-CART.

DETAILED DESCRIPTION:
PD1-CD19-CART is a kind of chimeric antigen T cell targeting CD19 with both CD19-CAR gene integration and also PD1 knockout by one-step gene-editing. After completion of study treatment, subject participation for this study will be followed up to 15 years post T cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Have the capacity to give informed consent;
2. ALL patients with the age between 18 and 70 years old;
3. Expected survival >3 moths;
4. With no severe heart and lung disease;
5. Previously confirmed diagnosis as CD19+ NHL within 6 months;
6. Hematological index as following, white blood cell (WBC)≥1.5×10^9/L，absolute neutrophil count (ANC) ≥0.8×10^9/L, Platelet count≥50×109/L, Hemoglobin (Hgb) ≥ 90mg/L, lymphocyte count≥ 0.4×10^9/L；
7. Blood biochemical index as no more than 1.5* ULN, including total bilirubin (TBIL), transglutaminase (AST), alanine aminotransferase (AST), Creatinine (SCr), Urea in patients with no tumor metastasis in liver and kidney; Blood biochemical index no more than 5* ULN in patients with tumor metastasis in liver and kidney;
8. With a stable cardiac function, the left ventricular ejection fraction (LVEF) ≥ 55%;
9. Virological tests were negative for EBV, CMV, HIV, TP and HCV; a negative HBV DNA test is acceptable if HBsAg is positive;
10. ECOG <2;
11. Relapsed or refractory (r/r) NHL including, Diffuse large B cell lymphoma(DLBCL, NOS), stage Ⅲ-Ⅳ;Primary mediastinal large B-cell lymphoma (PMBL), stage Ⅲ-Ⅳ; High grade B-cell lymphoma (HGBL), stage Ⅲ-Ⅳ; Mantle cell lymphoma (MCL), stage Ⅲ-Ⅳ; follicular lymphoma (FL), stage Ⅲ-Ⅳ and with aggression. r/r NHL defined as following, demonstrate disease that persists or relapse after achieving complete response (CR) after > 2 cycles of standard chemotherapy, or relapse after autologous hematopoietic stem cell transplantation (auto-HSCT), or not achieving CR after auto-HSCT.

Exclusion Criteria:

1. Pregnant or lactating women;
2. With a pregnancy plan in the next 2 years;
3. Prior treatment of anti-GVHD therapy;
4. Acceptance of allogeneic stem cell transplant (ASCT);
5. Isolated extramedullary relapse of ALL;
6. Severe mental disorders, active autoimmune diseases, active infectious diseases, severe cardiovascular diseases;
7. Partial prothrombin time or activated partial thromboplastin time or international standardized ratio > 1.5*ULN without anticoagulant treatment;
8. History of other type of maligant tumors;
9. Any circumstances that possibly increase the risk of subjects or interfere with study results, which judged by investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
MTD | up to 28 days after T cell infusion
  MTD will be determined based on DLTs observed during the first 28 days of study treatment.
RP2D | up to 28 days after T cell infusion
  RP2D will be determined based on MTD and efficiency during the first 28 days of study treatment.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Baseline up to 3 months after T cell infusion
  Proportion of patients in whom a response among complete response and partial response as defined by standard disease-specific criteria, will be observed.
Progress free survival (PFS) | Baseline up to 3 months after T cell infusion
  Assessed using modified Lugano classification response criteria for lymphoma (2014)

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, Prof, Principal Investigator — the First Affliated Hospital, Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu Y, Zu C, Zhang M, Wei G, Li W, Fu S, Hong R, Zhou L, Wu W, Cui J, Wang D, Du B, Liu M, Zhang J, Huang H. Safety and efficacy of CRISPR-based non-viral PD1 locus specifically integrated anti-CD19 CAR-T cells in patients with relapsed or refractory Non-Hodgkin's lymphoma: a first-in-human phase I study. EClinicalMedicine. 2023 May 18;60:102010. doi: 10.1016/j.eclinm.2023.102010. eCollection 2023 Jun. PMID 37251628
- [Derived] Zhou L, Fu W, Wu S, Xu K, Qiu L, Xu Y, Yan X, Zhang Q, Zhang M, Wang L, Hong R, Chang AH, Yu J, Fu S, Kong D, Li L, Wang Y, Li Z, Jiang H, Huang J, Liu Z, Su N, Wei G, Hu Y, Huang H. Derivation and validation of a novel score for early prediction of severe CRS after CAR-T therapy in haematological malignancy patients: A multi-centre study. Br J Haematol. 2023 Aug;202(3):517-524. doi: 10.1111/bjh.18873. Epub 2023 May 16. PMID 37192741
- [Derived] Zhang J, Hu Y, Yang J, Li W, Zhang M, Wang Q, Zhang L, Wei G, Tian Y, Zhao K, Chen A, Tan B, Cui J, Li D, Li Y, Qi Y, Wang D, Wu Y, Li D, Du B, Liu M, Huang H. Non-viral, specifically targeted CAR-T cells achieve high safety and efficacy in B-NHL. Nature. 2022 Sep;609(7926):369-374. doi: 10.1038/s41586-022-05140-y. Epub 2022 Aug 31. PMID 36045296
- [Derived] Golubovskaya V. CAR-T Cells Targeting Immune Checkpoint Pathway Players. Front Biosci (Landmark Ed). 2022 Apr 2;27(4):121. doi: 10.31083/j.fbl2704121. PMID 35468680